CLINICAL TRIAL: NCT05105958
Title: Tideglusib for the Treatment of Amyotrophic Lateral Sclerosis (TIDALS): a Randomized Placebo-controlled Phase II Trial
Brief Title: Tideglusib for the Treatment of Amyotrophic Lateral Sclerosis
Acronym: TIDALS
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Lausanne Hospitals (Other); University of Bern (Other); Cantonal Hospital of St. Gallen (Other); University Hospital, Geneva (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TIDALS_01
Record Dates: First submitted 2021-10-04; First posted 2021-11-03 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — tideglusib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tideglusib (Experimental): Patients receive 1000 mg Tideglusib once daily per os
  Interventions: Drug: Tideglusib
- Placebo (Placebo Comparator): Patients receive placebo matching Tideglusib 100 mg once daily per os
  Interventions: Drug: Tideglusib

INTERVENTIONS:
Drug: Tideglusib — 1000 mg/day per os

SUMMARY:
Amyotrophic lateral sclerosis (ALS) is a severe neurodegenerative condition, mainly characterized by progressive weakness and wasting of the limbs, the respiratory and bulbar muscles. Respiratory insufficiency leads to a fatal outcome after a mean diseases duration of only three to five years. The disease is characterized by pathological accumulations of a protein called TDP-43, which can be found large cortical and sub-cortical areas of post-mortem ALS brains.

No causal treatment for this condition is known to date, and there is a large unmet need to develop new strategies in order to halt or slow down its progression.

The aim of this study is to test the safety and tolerability of Tideglusib, a treatment that is already in clinical trials for other neuromuscular conditions, in patients with ALS. It is assumed that this drug may have a significant therapeutic benefit in this population due to his mode of action: In the ALS mouse model, Tideglusib decreases significantly the amount of accumulated TDP-43 proteins within the cells.

ELIGIBILITY:
Inclusion Criteria:

* Possible, probable (clinically or laboratory supported) or definite ALS according to the revised version of the El Escorial criteria
* Disease duration < 18 months
* Vital capacity of more than 60% of normal (defined as slow vital capacity, best of three measurements)
* Age more than 18 years
* On a stable dose of riluzole for at least four weeks or not taking riluzole
* On a stable dose of edaravone for at least four weeks or not taking edaravone
* Capable of thoroughly understanding all information given and giving full informed consent according to GCP

Exclusion Criteria:

* Previous participation in another clinical study within the preceding 12 weeks
* Proven SOD1- or FUS - mutation
* Tracheostomy or assisted ventilation of any type during the preceding three months
* Pregnancy or breast-feeding females
* Any medical condition known to have an association with motor neuron dysfunction which might confound or obscure the diagnosis of ALS
* Presence of any concomitant life-threatening disease or impairment likely to interfere with functional assessment
* Evidence of a major psychiatric disorder or clinically evident dementia precluding evaluation of symptoms
* Alcoholism
* Cardiovascular disorder/arrhythmia
* Impaired kidney function, defined as creatinine levels of 2.5 x upper limit of normal (ULN)
* Impaired liver function, defined as aspartate aminotransferase (AST) or alanine aminotransferase (ALT) of 3 x ULN
* Liable to be not cooperative or comply with trial requirements as assessed by the investigator, or unable to be reached in the case of emergency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Increase in Alanine Aminotransferase | 14 weeks
  Increase in Alanine Aminotransferase < 3x of Upper Limit of Normal

SECONDARY OUTCOMES:
Most common side effect | 14 weeks
  Occurence of diarrhea in less then 18 % of patients

OTHER OUTCOMES:
Exploratory outcome: clinical efficacy | 14 weeks
  Difference of decline in points on the Revised ALS Functional Rating Scale between the two study arms
Exploratory outcome: vital capacity | 14 weeks
  slow vital capacity in %

CONTACTS AND LOCATIONS:
Overall Officials: Annemarie Hübers, Principal Investigator — University Hospital, Geneva
Locations (5):
- Switzerland (5):
  - University Hospital Bern, Bern
  - University Hospital Geneva, Geneva
  - University Hospital Lausanne, Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No